CLINICAL TRIAL: NCT06490952
Title: Study on the Influencing Factors and the Pathways of Health Behavior in Patients After Heart Valve Replacement
Brief Title: Study of Health Behavior in Patients After Heart Valve Replacement： Longitudinal Studies
Status: Recruiting | Type: Observational
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024KY048
Record Dates: First submitted 2024-07-01; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-04

CONDITIONS: Heart Valve Diseases; Health Behavior; Postoperative Period
MeSH Terms: conditions — Heart Valve Diseases; Health Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigates the influencing factors and the pathways of health behavior in patients after heart valve replacement.

DETAILED DESCRIPTION:
Currently, the prevalence of heart valve disease is 2.0% to 13.2%, and heart valve replacement is the most important treatment to address heart valve disease. Heart valve replacement surgery is highly traumatic and risky, and the recovery of physiological, psychological, and social functions of postoperative patients is challenging, affecting the recovery process of patients. Healthy behavior is a lifestyle that can effectively reduce risk factors for adverse events and complications at the physiological, psychological, and social levels to slow disease progression, which can help promote patient recovery and improve prognosis. Therefore, this study investigates and analyzes the health behaviors of postoperative patients in different periods, explores their influencing factors and analyzes their pathways of action.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. VHD diagnosed by echocardiography;
3. Received HVR treatment;
4. able to communicate normally.

Exclusion Criteria:

1. Those with a conscious disorder or mental illness;
2. Those with severe organic diseases or comorbidities;
3. Those with cardiac function class IV;
4. Those who could not complete the questionnaire correctly independently or under the guidance of the researcher.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing postoperative heart valve replacement were selected for the study.
Sampling Method: Non-Probability Sample
Enrollment: 219 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Health behavior | At 1-2 days before discharge, at 1 month after discharge, at 3 month after discharge, at 6 month after discharge.
  A set of behavioral activities undertaken by an individual to promote or maintain health.

SECONDARY OUTCOMES:
Social support | At 1-2 days before discharge, at 1 month after discharge, at 3 month after discharge, at 6 month after discharge.
  Support received by an individual from within a social relationship.
Anxiety and depression | At 1-2 days before discharge, at 1 month after discharge, at 3 month after discharge, at 6 month after discharge.
  Measuring the psychological situation.
Self-efficacy | At 1-2 days before discharge, at 1 month after discharge, at 3 month after discharge, at 6 month after discharge.
  Measure the level of self-confidence.
Medication Literacy | At 1-2 days before discharge, at 1 month after discharge, at 3 month after discharge, at 6 month after discharge.
  Measuring medication-taking skills.

CONTACTS AND LOCATIONS:
Overall Officials: Yanjuan Lin, Study Chair — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No